CLINICAL TRIAL: NCT04616508
Title: Online Motor Control in People With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1358328-5
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Motor Control; Parkinson Disease
Keywords: motor control; Parkinson disease; motor learning
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral testing (Experimental)
  Interventions: Behavioral: motor control assessment

INTERVENTIONS:
Behavioral: motor control assessment — Basic science study of control of reaching movements

SUMMARY:
This study aims to better understand how people with Parkinson's control reaching movements. Specifically, we are asking how these individuals respond to different environmental perturbations. Testing includes reaching movements made within a virtual reality set-up.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disease, affecting approximately up to 10 million people worldwide and with 60,000 new cases diagnosed annually in the U.S. alone. Some of the most common signs and symptoms in individuals with PD are slowed and small movements and difficulty in movement initiation. The ability to correct movements online in response to environmental changes is an important part of daily living. Online movement corrections in reaching refer to the ability to smoothly change how and where you reach in response to a change in the environment. For example, one can adjust the position of the hand and arm when trying to catch a butterfly flying in the air. Generally speaking, online movement corrections can happen in response to visual perturbations (e.g., trying to catch a butterfly) or to force perturbations (e.g., someone knocks your hand while you're holding a coffee mug). Since individuals with PD have trouble with movements, it stands to reason that they may have problems with online movement corrections. Surprisingly, very little is known about online movement corrections in individuals with PD. The current evidence suggests that individuals with PD can make online movement corrections to small visual perturbations, but whether they can successfully respond to large visual perturbations is debatable. Furthermore, whether individuals with PD can make online movement corrections to force perturbations has not been studied. The aim of this project is to investigate if individuals with PD can make online movement corrections during reaching to visual and/or force perturbations. We will test both individuals with PD and age-matched healthy controls. They will perform reaching movements while visual or force perturbations are applied. We will use various perturbation strengths in order to test for potential differences in responses to small and large perturbations. Results from this study will provide new information on how individuals with PD make online movement corrections, and possibly provide insight to improving rehabilitation for PD.

ELIGIBILITY:
Inclusion criteria (all participants):

* Age 18-85 years
* Able to perform reaching movements of ~20 cm (8 inches)
* MMSE score ≥ 26/30
* Willing and able to attend all testing sessions

Inclusion criteria (PD group only):

* Diagnosis of idiopathic Parkinson's disease per self report
* Currently taking dopaminergic/dopamine agonist medication

Exclusion criteria (all participants):

* Any chronic or recent upper extremity musculoskeletal conditions that affects reaching
* Any neurological disorders other than Parkinson's disease (e.g., seizure disorders, closed head injuries with loss of consciousness greater than 15 minutes, CNS neoplasm, history of stroke)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
End-point errors | during intervention
  Euclidean distance from target to final hand position (units: cm); measurement derived from position data sampled at 1000 Hz
Reaction times | during intervention
  Time from visual target presentation to movement onset (units: ms); measurement derived from position data sampled at 1000 Hz
Movement times | during intervention
  Time from movement onset to movement end (units: ms); measurement derived from position data sampled at 1000 Hz

CONTACTS AND LOCATIONS:
Overall Officials: Hyosub Kim, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States